CLINICAL TRIAL: NCT06876948
Title: STUDY of NEUROLOGICAL COMPLICATIONS of LONG COVID-19 in CHILDREN and ADOLESCENTS; NEUROPSYCHIATRIC, ELECTROENCEPHALOGRAPHIC and NEURORADIOLOGICAL INVESTIGATIONS
Brief Title: NENCA Study on Neurological Complications of Long COVID-19 in Children and Adolescents; Neurophysiological, Electroencephalographic and Neuroradiological Investigation
Acronym: NENCA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, alessandro orsini, Alessandro Orsini, Azienda Ospedaliero, Universitaria Pisana
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: GR-2021-1237536; D65E2000350001 (Other Grant/Funding Number: Italian Ministry)
Record Dates: First submitted 2025-02-19; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Long Covid-19
Keywords: Covid-19
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19 | interventions — Electroencephalography; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Studio NENCA sulle complicanze neurologiche del Long Covid-19 nei bambini e negli adolescenti (Experimental): Patients are administered some psychological tests, if they are positive they move on to the next stage, otherwise the patients leave the practice. If they are positive, EEG, MRI and other psychological tests are also administered.
  Interventions: Diagnostic Test: Psychological tests, EEG, Magnetic Resonance

INTERVENTIONS:
Diagnostic Test: Psychological tests, EEG, Magnetic Resonance — Patients are administered some psychological tests, if they are positive they move on to the next stage, otherwise the patients leave the practice. If they are positive, EEG, MRI and other psychological tests are also administered.

SUMMARY:
The study seeks to investigate the neurological effects caused by Covid-19 in children and adolescents in the 6-16 age group. To do this, neuropsychological scales, an EEG and an MRI were used.

ELIGIBILITY:
Inclusion Criteria:

* Age between 6 years and 16 years and 11 months
* Symptomatology compatible with long neurological COVID, specifically: persistence or appearance of new neurological signs/symptoms (e.g. fatigue, headache, sleep disturbance, cognitive dysfunction, memory difficulties, emotional or mood disorders, vertigo cognitive dysfunction, memory difficulties, emotional or mood disorders, dizziness, dysautonomia, movement disorders movement disorders, ataxia, tremor, epilepsy, muscle weakness, myalgia, hyposmia, hypogeusia hearing loss or tinnitus and/or sensorimotor deficits such as hypoesthesia, dysesthesia) after three months after established SARS-CoV-2 infection, as well as persistence of these symptoms for at least two months, in the absence of a clear aetiology.
* Signature of the appropriate Informed Consent by caregiver(s) and patient(s)

Exclusion Criteria:

* Poor knowledge of the Italian language or other limitation of verbal communication that compromises the subject's ability to perform neuropsychological tests
* Need for sedation to perform brain MRI 7 Tesla
* Neurological or neuropsychiatric disorder diagnosed prior to COVID-19 diagnosis
* Caregiver's failure to sign consent

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2023-03-29 (Actual); Primary Completion 2025-03-29 (Estimated); Study Completion 2026-04-28 (Estimated)

PRIMARY OUTCOMES:
Changes in cognitive and neuropsychological functions in children and adolescents with Long COVID between T0 and T1. | Test administration at the time of diagnosis of Long COVID (T0) and follow-up after 6-9 months (T1).
  Assessment of cognitive, neuropsychological and adaptive skills in children and adolescents with Long COVID by means of standardised tests (WISC-IV, CPT3, NEPSY II, BRIEF-2, Vineland Adaptive Behavior Scales). The tests measure attention, memory, executive functions, intellectual-adaptive functioning and quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Universitaria Pisana, Pisa, PI, Italy

IPD SHARING:
Plan to Share IPD: Yes